CLINICAL TRIAL: NCT01264913
Title: Cardiometabolic Risk of ShiftWork: Sleep Loss vs.Circadian Disruption
Brief Title: Cardiometabolic Risk of Shiftwork
Acronym: SW
Status: Terminated | Type: Observational
Why Stopped: impossible to retain participants in 3-year longitudinal study
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 09-049-A
Record Dates: First submitted 2010-12-13; First posted 2010-12-22 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Sleep Deprivation; Circadian Dysregulation; Shift-Work Sleep Disorder
MeSH Terms: conditions — Sleep Deprivation; Chronobiology Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Shift Workers
  Interventions: Behavioral: sleep extension & circadian alignment
- Day Workers
  Interventions: Behavioral: sleep extension & circadian alignment

INTERVENTIONS:
Behavioral: sleep extension & circadian alignment — Both groups of workers will undergo a 1-week period of fixed bedtimes, light-dark cycles and mealtimes in the laboratory to pay the sleep debt and align the circadian system
  Other Names: SWI intervention

SUMMARY:
The overall goal of the present application is to test the hypothesis that shift workers, who are chronically exposed to circadian misalignment and sleep loss, have a higher cardio-metabolic risk than day workers, and that the accumulated sleep debt and the degree of circadian misalignment both predict their elevated cardio-metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Day workers and shift workers at the University of Chicago, University of Chicago Medical Center, or another Chicago area medical center who have maintained their work schedule (at least 30 hours/week) for at least 6 months.
* Individuals who have been shift workers for less than 10 years; body mass index <40 kg/m2;
* No major illness
* No history of psychiatric, endocrine, cardiac or sleep disorders
* Those with hypertension or dyslipidemia will be included if these conditions are controlled by a stable treatment.
* Women taking oral contraceptive or hormonal replacement therapy will be included only if they plan to stay on a stable regimen throughout the study.
* Age must be between 18 and 50 years

Exclusion Criteria:

* Individuals who have worked at the University of Chicago, University of Chicago Medical Center, or another Chicago area medical center in their current position for less than 6 months.
* Individuals who have been shift workers for more than 10 years
* BMI>40 kg/m2
* Individuals with a major illness (e.g. diabetes, sleep disorder)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will enroll 44-46 regular day workers (work hours between 7:00 a.m. and 7:00 p.m. on all work days) and 44-46 shift workers on rotating schedules (changing shift at lease once a week and having work hours between 7:00 p.m. and 7:00 a.m. on at least 10 days per month). Both groups of subjects will work at least 30 hours per week at the University of Chicago, University of Chicago Medical Center, or other Chicago area medical center and have maintained their work schedule for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States